CLINICAL TRIAL: NCT02049125
Title: Urinary Biomarker NGAL in Decompensated Cirrhosis: Early Prediction of AKI and of Treatment Response
Brief Title: Study of Accuracy of NGAL, a Renal Injury Biomarker, in Patients With Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Federal University of Espirito Santo (Other); Hospital de Base (Other); University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Alberto Queiroz Farias, Associate Professor of Medicine School of University of Sao Paulo, University of Sao Paulo
Other Study IDs: NGAL01
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Acute Kidney Injury; Hepatorenal Syndrome
Keywords: NGAL; Acute kidney injury; Cirrhosis; Hepatorenal syndrome
MeSH Terms: conditions — Acute Kidney Injury; Hepatorenal Syndrome; Fibrosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will store samples of urine and serum frozen at -80oC.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No AKI: Patients with cirrhosis admitted to hospital with bacterial infection with initial serum creatinine below 1.5mg/dL.
- AKI and Infection: Patients with cirrhosis admitted to hospital with bacterial infection and initial serum creatinine above 1.5mg/dL.
- AKI with No Infection: Patients with cirrhosis admitted to hospital with initial serum creatinine above 1.5mg/dL without bacterial infection.

SUMMARY:
The purpose of this study is to test the accuracy of urinary neutrophil-gelatinase associated lipocalin (NGAL) and other biomarkers (plasma renin, norepinephrine) to predict acute kidney injury (AKI) development in patients with cirrhosis and bacterial infection and to predict response to AKI treatment with albumin and albumin with terlipressin in patients with suspected hepatorenal syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis diagnosis by liver biopsy or combination of clinical, laboratorial, endoscopic and imagenological data;
* Presence of ascites and/or hepatic hydrothorax;
* Age over 18 years old;
* Diagnosis of bacterial infection (including spontaneous bacterial peritonitis and others) with or without acute kidney injury (defined as a serum creatinine above 1.5mg/dL at admission) or acute kidney injury without bacterial infection;
* Agreement to participate in the study, registered by informed consent;

Exclusion Criteria:

* Serious comorbidities (functional class IV heart failure, O2 dependent chronic obstructive pulmonary disease, advanced cancer);
* Shock, as defined by American College of Chest Physicians;
* Chronic kidney disease with serum creatinine persistently above 1.5mg/dL in the previous 6 months and/or with sonographic findings of chronic nephropathy;
* Intrinsic nephropathy with hematuria over 50 red cells/high power field and dysmorphic erythrocyte and/or proteinuria over 500mg/24h;
* Use of nephrotoxic drugs in the previous 30 days;
* Dialysis prior to study inclusion;
* Previous solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include cirrhotic patients admitted to hospitals participating centers with AKI and/or bacterial infection.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy of NGAL to predict no response to albumin expansion | One day after albumin expansion (day 3)
  We will build a receiver-operating curve and calculate the area under the curve to determine the accuracy of NGAL to predict no response to albumin expansion. No response will be defined as an absence of a drop of serum creatinine to a final value below 1.5mg/dL in the day after the end of albumin expansion. Albumin will be administrated as International Ascites Club recommendations, i.e. in the dose of 1g/kg/day for 2 days in patients with suspected hepatorenal syndrome.

SECONDARY OUTCOMES:
Accuracy of urinary NGAL and other biomarkers to predict no response to hepatorenal syndrome treatment | Treatment period (maximum of 14 days)
  We will test the accuracy of urinary NGAL and other biomarkers to predict no response to hepatorenal syndrome treatment. No response to treatment will be defined as a final value of serum creatinine above 1.5mg/dL after the end of treatment with terlipressin plus albumin. The treatment will be conducted according to International Ascites Club recommendations.
Accuracy of urinary NGAL and other biomarkers to predict development and progression of acute kidney injury (AKI) in patients with bacterial infection | During antibiotic therapy and during hospital stay
  We will test the accuracy of urinary NGAL and other biomarkers to predict AKI development and progression during antibiotic therapy and during hospital stay in patients with bacterial infection. AKI will be defined by ICA-AKI criteria.
Predictors of mortality | In-hospital, 30 days and 90 days
  We will test clinical and laboratorial data relationship with in-hospital, 30 days and 90 days mortality in a univariate analysis. Associated variables will be tested in a multivariate analysis.
Urinary NGAL as a predictor of adverse events of AKI treatment in cirrhosis | During treatment period
  We will build a receiver-operating curve and calculate the area under the curve to determine the accuracy of urinary NGAL to predict adverse events during AKI treatment with albumin alone or in combination with terlipressin. We will also calculate the best cut-off value based on the receiver-operating curve.
Accuracy of other biomarkers to predict no response to albumin expansion | One day after albumin expansion (day 3)
  We will test the accuracy of other biomarkers to predict no response to albumin expansion. No response will be defined as an absence of a drop of serum creatinine to a final value below 1.5mg/dL in the day after the end of albumin expansion. Albumin will be administrated as International Ascites Club recommendations, i.e. in the dose of 1g/kg/day for 2 days in patients with suspected hepatorenal syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Q Farias, Associate professor, Study Chair — University of Sao Paulo
Locations (4):
- Brazil (4):
  - Federal University of Espirito Santo, Vitória, Espírito Santo
  - Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - University of Campinas, Campinas, São Paulo
  - University of Sao Paulo, São Paulo, São Paulo